CLINICAL TRIAL: NCT00421798
Title: Rapid Characterization of Mycobacteria and Drug Resistance In Paucibacillary TB
Brief Title: Rapid Characterization of Paucibacillary TB Along Tex/Mex Border
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Blanca I Restrepo, PhD - Principal Investigator, UT Health Science Center at Houston -School of Public Health
Other Study IDs: 06-0042 transfer from DMID; NCT00763854 (obsolete NCT alias)
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Mycobacterium Tuberculosis
Keywords: tuberculosis, paucibacillary, mycobacteria, Mexico, Colombia
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood from participants will be collected, and DNA extracted from white blood cells. These are expected to also contain DNA from M. tuberculosis- that will be the research question
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will test a method of detecting tuberculosis-causing bacteria that are resistant to current medication treatments. Blood samples will be collected from patients from 3 sites and 3 mainly Hispanic populations in Texas, Mexico, and Colombia. Up to 780 males and females, ages 18-85 years, will participate. The study population will consist of 390 people with any of 3 forms of tuberculosis (TB) and 390 people who are either healthy or with a disease initially thought to be one of these 3 forms of TB but then ruled out. Volunteers will only be contacted, invited to participate and interviewed at the beginning of their evaluation for possible TB.The study team will follow up with the health department to determine if the volunteer was indeed diagnosed with TB, and with the laboratory to determine the results of TB tests at diagnosis and during the course of treatment.

DETAILED DESCRIPTION:
Global challenges to tuberculosis (TB) control are multidrug resistance TB (MDR-TB) and the increased susceptibility of populations such as elderly, those with HIV infection, type 2 diabetes and other immunosuppressive chronic diseases. The first primary study objective is to examine the potential of the investigators' new DNA extraction/qPCR protocol as a non-invasive tool to study pathogenesis in a range of paucibacillary specimens. The investigators will evaluate their DNA extraction/qPCR assays prospectively in specimens from patients with paucibacillary TB, including extra-pulmonary TB (EPTB) and smear-negative pulmonary TB. Investigators will determine the number of mycobacterial genomes, presence of intact mycobacteria, and precise location within plasma, PBMCs or PMNs in blood, or other fluid or cells in a range of specimens. The second primary study objective is to standardize and validate a qPCR assay for early detection of Mycobacterium tuberculosis (MTB) drug resistance directly from specimens. The investigators will further establish the feasibility of using this highly sensitive assay to determine the ratio of Rifampin (RIF)-resistant to RIF-susceptible bacteria in a given specimen. The investigators will adapt a simple and effective method, similar to their qPCR technology, for detection of mutations in the rpoB gene. MTB-positive specimens, identified by either qPCR or direct smear, will be screened for RIF resistance using molecular beacons as probes in qPCR. The concordance between the molecular beacon-qPCR assays and resistance phenotype from culture will be established. The investigators will then utilize the capacity of qPCR to quantitate ratios of RIF-resistant to -sensitive mycobacteria in a clinical specimen. The investigators hypothesize that current assays are limited to indicating "presence" of drug susceptibility but in the patient the situation is more complex, with dynamic mixtures of resistant and sensitive bacteria, depending on local exposure to drugs. Developing a tool that detects minor populations of drug-resistance cells will open new avenues of investigation to help understand development of resistance and treatment failures. Primary study outcomes include: anticipation that the qPCR in blood WBCs will provide substantially improved sensitivity and precision (mycobacterial species information) in the diagnosis of paucibacillary TB, specifically tuberculous lymphadenitis, pleural TB and smear-negative (early) pulmonary TB, when compared with standard microbiological and clinical diagnosis; anticipation that molecular beacon-qPCR will predict RIF-resistance with 100% sensitivity and at least 86% sensitivity in their study site, providing a new tool for early suspicion of MDR, and hence, prompt modification in the treatment schedule of the patient; and investigators will learn about the biology of emergence of RIF resistance in a population of mycobacteria from serial patient specimens. Specimens will be collected from patients from 3 sites, all with predominantly Hispanic populations, located in South Texas, adjacent northeast Mexico, and Colombia. A maximum of 780 males and females, ages 18-85 years, will be recruited. The study population will consist of 390 people with tuberculosis (62 with TB lymphadenitis, and at most 164 with pleural TB and 164 with smear-negative pulmonary TB) and 390 controls (either healthy controls or with a disease initially thought to be one of the three forms of TB described for cases, but then ruled out). Subjects will have 1 study related visit. Patients will only be contacted, invited to participate and interviewed at the beginning of their evaluation for possible TB. The study team will follow-up with the health department to determine if the patient was indeed diagnosed with TB, and with the laboratory to determine the results of serial direct smear, culture and sensitivity at diagnosis and during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

For Cases and Controls:

* Informed consent obtained and signed
* Older than 18 years of age, up to 85 years of age

Unique to Cases:

-Suspicion of smear-negative pulmonary tuberculosis, lymphatic tuberculosis or pleural tuberculosis

Unique to Controls:

* Initial suspicion of tuberculosis (as described under cases) but diagnosis eventually ruled out through further testing
* Patient with another pathology where specimen similar to that collected for the cases is also obtained, and leftover material is available for this study; example- lymph node biopsy from a patient with cancer

Exclusion Criteria:

* Patient having received more than 14 days of anti-mycobacterial treatment
* Less than 18 years old
* Prisoner or jail inmate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Studies will be conducted in the population from the TExas-Mexico border, and in Colombia. Participants are TB suspects, or controls.
Sampling Method: Non-Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Restrepo, PhD, Principal Investigator — UT Health Science Center at Houston -School of Public Health
Locations (3):
- The University of Texas at Brownsville, Brownsville, Texas, United States
- Corporacion para Investigaciones Biologicas de Medellin, Medellín, Colombia
- Jurisdicción Sanitaria III Matamoros, Matamoros, Mexico